CLINICAL TRIAL: NCT04465487
Title: A Phase 1 Study of REGN6569, an Anti-GITR mAb, With Cemiplimab in Patients With Advanced Solid Tumor Malignancies
Brief Title: Study of REGN6569 and Cemiplimab in Adult Patients With Advanced Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R6569-ONC-1933; 2020-000075-20 (EudraCT Number)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Unselected solid tumors dose escalation; HNSCC dose expansion; Advanced stage solid tumor malignancy; Unresectable; Metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): REGN6569 lead-in, then combo therapy
  Interventions: Drug: REGN6569; Drug: Cemiplimab
- Dose Expansion (Experimental): Randomized 1:1 between cohorts Cohort 1: Concurrent start of REGN6569 + cemiplimab Cohort 2: REGN6569 lead-in, then combo therapy
  Interventions: Drug: REGN6569; Drug: Cemiplimab

INTERVENTIONS:
Drug: REGN6569 — Administered by intravenous (IV) infusion
Drug: Cemiplimab — Administered by IV infusion
  Other Names: REGN2810; Libtayo

SUMMARY:
There are two main goals of this study: The first is to find the highest safe dose of REGN6569 when given with cemiplimab. The second is to get some initial information about how well the REGN6569 in combination with cemiplimab may help shrink certain types of cancer.

The study is also looking at:

* Side effects that may be experienced by people taking REGN6569 alone and with cemiplimab
* How REGN6569 and cemiplimab work in the body
* How much REGN6569 and cemiplimab is in your blood
* To see if REGN6569 can lower the number of Treg cells in tumors
* To see if REGN6569 and cemiplimab can shrink tumors when given together

ELIGIBILITY:
Key Inclusion Criteria:

1. Dose escalation cohorts: Advanced stage (unresectable or metastatic) solid tumor malignancy, confirmed histologically or cytologically as defined in the protocol
2. Dose expansion cohorts: Advanced stage (unresectable or metastatic) head and neck squamous cell carcinoma (HNSCC), confirmed histologically or cytologically. Patients must have evidence of progression on anti-Programmed death-1 (receptor)/Programmed death ligand 1 (PD-1/PD-L1) blockade either as monotherapy or in combination with other therapies, as defined in the protocol
3. Mandatory biopsies: Able and willing to provide tumor tissue at baseline and while on treatment, with at least 1 soft tissue lesion amenable to biopsy by ultrasound or computed tomography (CT)-guided biopsy or under direct visualization as defined in the protocol

Key Exclusion Criteria:

1. Has previously received GITR-targeted therapy
2. Has received any previous systemic biologic therapy within 5 half-lives of first dose of study therapy as defined in the protocol
3. Has any condition that requires ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 14 days prior to the first dose of study therapy
4. Has ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments as defined in the protocol
5. Has a known history of, or any evidence of, interstitial lung disease, or active, non-infectious pneumonitis in the past 5 years. A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥6 months prior to first dose of study therapy
6. Has uncontrolled infection with human immunodeficiency virus, hepatitis B or hepatitis C infection, or diagnosis of immunodeficiency
7. Has received a live vaccine within 4 weeks of planned start of study medication. For dose escalation only: Has received a COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study.
8. Has had prior allogeneic stem cell transplantation or received organ transplants at any time, or autologous stem cell transplantation
9. Has a history of malignancy within 2 years of date of first planned dose on study as defined in the protocol

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limited toxicities (DLTs) | Up to 42 days
  Dose escalation period
Incidence and severity of treatment emergent adverse events(TEAEs) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation period
Incidence and severity of adverse events of special interest (AESIs) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation period
Incidence and severity of serious adverse events (SAEs) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation period
Incidence and severity of grade ≥3 laboratory abnormalities | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation period
Objective response rate (ORR) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose expansion period
Characterize percentage change in intratumoral glucocorticoid-induced tumor necrosis factor receptor-Related (GITR)+ Treg density | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose expansion period

SECONDARY OUTCOMES:
ORR | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation period
Disease control rate (DCR) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Duration of Response (DOR) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Progression-free Survival (PFS) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Overall survival (OS) | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Drug concentrations of REGN6569 in serum | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Drug concentrations of cemiplimab in serum | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Immunogenicity as measured by anti-drug antibodies (ADA) to REGN6569 | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods
Immunogenicity as measured by anti-drug antibodies (ADA) to cemiplimab | Up to 90 days after the last dose of REGN6569 and/or cemiplimab, whichever is administered last, an average of approximately 30 months
  Dose escalation and expansion periods

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (4):
  - Angeles Clinic and Research Institute - Clinic/Outpatient Facility, Los Angeles, California
  - H.Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - START South Texas Accelerated Research Therapeutics, Grand Rapids, Michigan
- Spain (6):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/